CLINICAL TRIAL: NCT00467584
Title: Aspirin for Treatment of Multiple Sclerosis-Related Fatigue
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis indicated treatment unlikely effective;slow recruitment
Sponsor: Mayo Clinic (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Dean Wingerchuk, Professor of Neurology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-004850
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Aspirin (Active Comparator): High Dose Aspirin; 1300 milligrams of aspirin per day, taken by mouth as two tablets, twice per day for 8 weeks
  Interventions: Drug: High Dose Aspirin (1300 mg/day)
- Low Dose Aspirin (Active Comparator): Low Dose Aspirin; 162 milligrams of aspirin per day (the equivalent of 2 baby aspirin tablets) taken by mouth as two tablets, twice a day in the morning and at noon for 8 weeks
  Interventions: Drug: Low Dose Aspirin (162 mg/day)
- Placebo (Placebo Comparator): Placebo tablets, matching the active aspirin tablets in appearance, taken by mouth twice per day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High Dose Aspirin (1300 mg/day) — 1300 milligrams per day (the equivalent of 4 regular aspirin tablets) taken by mouth as two tablets, twice a day in the morning and at noon for 8 weeks
  Other Names: acetylsalicylic acid; ASA; Aspirin
  Arms: High Dose Aspirin
Drug: Low Dose Aspirin (162 mg/day) — 162 milligrams per day (the equivalent of 2 baby aspirin tablets) taken by mouth as two tablets, twice a day in the morning and at noon for 8 weeks
  Other Names: acetylsalicylic acid; ASA; Aspirin
  Arms: Low Dose Aspirin
Drug: Placebo — Placebo tablets matching the active aspirin tablets in appearance, taken as two tablets, twice per day for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether aspirin is effective for treatment of fatigue caused by multiple sclerosis (MS).

DETAILED DESCRIPTION:
Fatigue is the most common symptom of multiple sclerosis (MS), affecting up to 90% of people with the disease. MS-related fatigue can be disabling even when other features of MS are mild. It can interfere with physical activity, memory and thinking, social and family activities, and ability to work. Initial treatment consists of energy conservation techniques such as rest periods or naps but when these approaches fail doctors usually recommend a trial of medications. Amantadine, modafinil, and other stimulants are commonly used but help only about half of those who try them. It is unlikely that these drugs directly affect the cause of MS-related fatigue.

It has been difficult to develop new drug therapies for MS-related fatigue because we do not fully understand its causes and do not have precise ways to measure it. We rely on a person's self-report about their fatigue but individuals experience and report fatigue differently. Recent research has shown that some fatigue aspects, such as difficulty maintaining mental concentration ("cognitive fatigue") and physical activity ("motor fatigue"), can be measured more precisely and require further study.

We recently reported results from a study showing that people taking the equivalent of four regular aspirin tablets (1300 mg) daily had reduced MS-related fatigue compared with placebo (sugar pill). The current proposal will attempt to confirm the benefit of aspirin in a larger group of people and to determine if the benefit is related to inflammation. One hundred and thirty-five people with MS-related fatigue will participate at MS clinics at three Mayo Clinic sites. Participants will complete questionnaires that ask about the severity and impact of their fatigue, memory testing to assess cognitive fatigue, and have blood testing to measure markers of inflammation. At the Arizona site, participants will also do strength testing in a motor laboratory to assess motor fatigue. After obtaining two separate baseline evaluations, the participants will be randomly assigned treatment such that one-third will receive 1300 mg per day of aspirin, one-third will receive 162 mg per day of aspirin and one-third will receive a matching placebo. All participants will then return to the clinic on two more occasions over the next eight weeks to repeat the questionnaires, memory and strength testing, blood tests, and report any side-effects. At the end of the study, the results of one of the fatigue questionnaires will be analyzed to determine if aspirin significantly improved fatigue compared with the placebo. The results of other questionnaires and the memory and strength testing will be analyzed as supportive evidence.

If this study is successful, it will provide strong scientific evidence that aspirin helps MS-related fatigue. It will add an important new option for treatment of all MS patients that is also familiar, inexpensive, and has a good long-term safety record. At the same time, it will allow us to better understand the causes of MS-related fatigue and how to measure it more precisely. This information will be extremely useful for development of other therapies in the future.

ELIGIBILITY:
Inclusion criteria:

* Confirmed relapsing-remitting or secondary progressive multiple sclerosis,
* Ambulatory for distance of at least 100 meters without gait assistance,
* Persistent fatigue for at least 8 weeks that is not attributable to causes other than MS, and
* Will be able to complete questionnaires and cognitive testing.

Exclusion criteria:

1. Other evident causes for fatigue:

   * Untreated depression or screening Center for Epidemiologic Studies Depression (CES-D) scale greater than 28
   * Significant cognitive impairment (Baseline Short Test of Mental Status score of less than 29/38)
   * Narcolepsy, uncontrolled sleep apnea, or other primary sleep disorder judged to be likely a major contributor to fatigue
   * Screening Epsworth Sleepiness Scale score greater than 15
   * Uncontrolled hypothyroidism or anemia
   * Other medical illness judged by the investigator to affect the participant's fatigue complaints including current viral, bacterial, mycobacterial, or fungal infection
2. MS Disease Activity and Treatment:

   * Clinical exacerbations within 2 weeks prior to screening visit
   * Corticosteroid use within 4 weeks prior to screening visit
   * Beta-interferon, glatiramer acetate, immunosuppressant drugs (mitoxantrone, azathioprine, etc.) are permitted if a stable dose has been used for greater than or equal to 4 weeks and there is no temporal association of drug administration with perceived fatigue; elective on-study dose/regimen changes are not permitted
3. Current or Recent Fatigue Therapy and Other Medications:

   * Use of more than two doses of ASA (aspirin) greater than 81 mg/d within 2 weeks of screening visit
   * Use of MS fatigue medications within 2 weeks of screening visit (including amantadine or Central Nervous System stimulants such as modafinil, methylphenidate, and pemoline)
   * Symptomatic medications (antidepressants, anti-spasticity agents, non-narcotic analgesics) are permitted if a stable dose has been used for >4 weeks prior to screening for antidepressants and >2 weeks prior to screening for other symptomatic therapies and there is no temporal association of drug administration with perceived fatigue; elective on-study dose changes are not permitted.
   * Current use of acetazolamide, antiplatelet agents or anticoagulants, COX-2 inhibitors, methotrexate, oral hypoglycemic medications
4. Medical Contraindications to ASA use:

   * Allergy to ASA or Non-Steroidal Anti-Inflammatory drugs
   * Syndrome of asthma, rhinitis and nasal polyps
   * History of confirmed peptic ulcer or gastrointestinal or severe gynecological bleeding
5. General Health Concerns:

   * Significant uncontrolled disease of cardiovascular, pulmonary, hepatic, renal, endocrine, rheumatological, neurological, gynecological, or gastrointestinal systems
   * Pregnancy or unwillingness to utilize contraception
   * History of alcohol or drug abuse within 6 months of screening or current alcohol intake >3 drinks/day
6. Laboratory Exclusions (available values obtained within 8 weeks prior to screening visit are acceptable for all except the pregnancy test)

   * Positive pregnancy test
   * Hemoglobin less than 11.0 g/dL (women) or 13.0 g/dL (men)
   * Platelet count < 120, 000/μL
   * Serum creatinine level > 1.4 mg/dL (women) or 1.6 mg/dL (men)
   * Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) level greater than 2.5 times the upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean M. Wingerchuk, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Multiple Sclerosis were recruited from three Mayo Clinic sites (Arizona, Minnesota and Florida) beginning in July, 2007.
Period: Overall Study
Arm/Group | High Dose Aspirin | Low Dose Aspirin | Placebo
Started | 21 | 20 | 21
Completed | 17 | 15 | 20
Not Completed | 4 | 5 | 1
Not completed — Withdrawal by Subject | 4 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Aspirin: Low Dose Aspirin; 162 milligrams of aspirin per day taken by mouth as two tablets, twice per day for 8 weeks
- Total: Total of all reporting groups
Arm/Group | High Dose Aspirin | Low Dose Aspirin | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 21 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.6) | 47.0 (10.3) | 47.4 (8.0) | 47.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 18 | 50
  Male | 4 | 5 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: Modified Fatigue Impact Scale Score
Description: The Modified Fatigue Impact Scale is a list of 21 statements describing how fatigue may affect a person's functioning. Answers ranging from 0 (Never) to 4 (Almost always) were provided by the study subjects for the prior 4 week period. A total score was tallied from a possible 0 (no fatigue impact) to 84 (almost always impacted by fatigue). A lower total score indicates less fatigue-related impact while a higher total score indicates greater fatigue-related impact on a subject's functioning.
Time Frame: Baseline, 8 weeks
Population: 62 patients were randomized; of these, 6 did not receive the intervention and an additional 4 discontinued without providing followup data. Therefore 52 were included in the analysis. The Wk 4 MFIS score was used if the subject withdrew prior to Wk 8. 1 subject each in the High Dose and Placebo groups provided MFIS data at Wk 4 but not Wk 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose Aspirin | Low Dose Aspirin | Placebo
Number analyzed (Participants) | 17 | 15 | 20
units on a scale
  MFIS Total Score at Baseline | 48 (13) | 50 (15) | 49 (13)
  MFIS Total Score at 8 Weeks | 37 (11) | 45 (17) | 44 (13)
  Change in MFIS Total Score | -11.4 (13.9) | -5.1 (15.7) | -5.5 (9.8)

ADVERSE EVENTS:
Time Frame: Baseline to 8 weeks
Arm/Group | High Dose Aspirin | Low Dose Aspirin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 5/17 | 0/15 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Aspirin (N=17) | Low Dose Aspirin (N=15) | Placebo (N=20)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Bladder infection
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nevus removal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Mole removed
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No